CLINICAL TRIAL: NCT05573906
Title: Augmenting the Efficacy of Benzodiazepine Taper With Telehealth-Delivered Cognitive Behavioral Therapy for Anxiety Disorders in Patients Using Prescription Opioids
Brief Title: Benzodiazepine Taper With Cognitive Behavioral Therapy in Patients Using Prescription Opioids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Boston University (Other)
Responsible Party: Principal Investigator, Kate Taylor, Associate Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB#22-001451; R21DA053394 (NIH); NCT05845606 (obsolete NCT alias)
Record Dates: First submitted 2022-10-05; First posted 2022-10-10 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive behavioral therapy for anxiety plus benzodiazepine taper (Experimental): 11 sessions of individual therapy consisting of exposure-based cognitive behavioral therapy that is designed specifically for assisting with benzodiazepine taper. This will be added to a gentle, 12-week benzodiazepine taper. CBT will be initiated for two sessions prior to the benzodiazepine taper initiation.
  Interventions: Combination Product: Cognitive behavioral therapy for anxiety plus benzodiazepine taper
- Health education control plus benzodiazepine taper (Active Comparator): 11 sessions of individual therapy control consisting of psychoeducational topics related to health and well-being, along with the gentle, 12-week benzodiazepine taper.
  Interventions: Combination Product: Health education control plus benzodiazepine taper

INTERVENTIONS:
Combination Product: Cognitive behavioral therapy for anxiety plus benzodiazepine taper — 11 sessions of individual therapy consisting of exposure-based cognitive behavioral therapy that is designed specifically for assisting with benzodiazepine taper. This will be added to a gentle, 12-week benzodiazepine taper. CBT will be initiated for two sessions prior to the benzodiazepine taper initiation.
  Arms: Cognitive behavioral therapy for anxiety plus benzodiazepine taper
Combination Product: Health education control plus benzodiazepine taper — 11 sessions of individual therapy control consisting of psychoeducational topics related to health and well-being, along with the gentle, 12-week benzodiazepine taper.
  Arms: Health education control plus benzodiazepine taper

SUMMARY:
Taking prescription opioids for pain together with benzodiazepines for the treatment of anxiety disorders is not recommended by the U.S. Food and Drug Administration (FDA) because of the elevated risk of serious complications, including fatal overdose. However, this concurrent prescription use continues to be prevalent, likely due to the high comorbidity between pain and anxiety disorders. Efforts are urgently needed to reduce benzodiazepine use among patients taking opioids. Cognitive behavioral therapy (CBT) is a first-line treatment for anxiety disorders, and represents a safer and more effective treatment for anxiety disorders compared to benzodiazepines. The proposed study aims to make minor adaptations to a CBT protocol to facilitate benzodiazepine tapering and to then conduct a 2-arm randomized clinical trial with primary care patients who receive benzodiazepine and opioid prescriptions. Participants will be randomized to receive a telehealth-delivered intervention consisting of a gentle, 12-week benzodiazepine taper (BZT) with either CBT or a health education control (HE). Participants will be assessed at baseline, several points throughout treatment, at post-treatment, and at a 2-month follow-up assessment on benzodiazepine use, opioid use, and anxiety symptoms. Should CBT + BZT outperform HE + BZT, this intervention could make a significant impact by reducing major consequences of concurrent use of opioids and benzodiazepines, including mortality.

ELIGIBILITY:
Inclusion Criteria:

* taking prescribed BZs for at least 3 months prior to baseline and have a positive UDS for BZs at baseline
* currently experiencing significant distress or impairment due to their anxiety symptoms (i.e., score ≥ 6 on the OASIS during screening
* have been prescribed opioids for at least 3 months for pain management and have a positive UDS for prescribed opioids at baseline
* are between 18-85 years old
* are fluent in English
* have access to a digital device with internet access for telehealth
* are willing to reduce BZ use.

Exclusion Criteria:

* pregnancy
* psychiatric symptoms requiring a higher level of care (i.e., severe suicidality, manic or psychotic symptoms not stabilized on medication)
* presence of any SUD other than tobacco use disorder, OUD (co-occurring with pain condition) or sedative/hypnotic use disorder)
* medical conditions that require ongoing treatment with benzodiazepines (e.g., certain seizure disorders)
* use of drugs other than BZs and opioids in the past 30 days (as indicated by UDS and self-report), with the exception of intermittent cannabis use (not meeting criteria for CUD) and use of alcohol above at-risk drinking cutoffs per US Dietary Guidelines
* marked cognitive impairment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Adherence | at week 15
  number of sessions attended
Treatment Satisfaction Questionnaire | at week 15
  This measure will be used to assess patient satisfaction and acceptability with the interventions.
Timeline Followback (change in benzodiazepine and opioid use and dose) | Baseline, weeks 1-14, post-treatment (week 15), and 2 months from week 15
  Timeline Followback (TLFB) will be used to assess BZ use and dose, opioid use and dose, and other substance use (and frequency and quantity). BZ dose at each assessment period will be assessed via self-report. Data will be gathered with the Timeline Followback (TLFB62), and facilitated by a dose diary card that patients will be given to track substance use (i.e., days of use of each drug including BZs) and dose of BZ on each day of BZ use. The diary card will only be used as a tool for participant recall during the TLFB administration, and will not be collected as data. TLFB administration will also be enhanced by asking patients to show their BZ pill bottles TLFB will be used to document self-reported use of substances for each day since the last TLFB assessment during the acute treatment phase (i.e., past 7 days during weekly study visits) and in the past 30 days for baseline, post-treatment, and follow-up (past month)
Depression Anxiety and Stress Scale (change in scores over time) | Baseline, weeks 1-14, post-treatment (week 15), and 2 months from week 15
  Primary outcome measure to assess anxiety symptoms (anxiety subscale will be primary; depression and stress subscales will be examined as secondary)

SECONDARY OUTCOMES:
Urine Drug Screen (UDS) | Baseline, post-treatment (week 15), and 2 months from week 15
  UDS panel will include benzodiazepines, opiates, buprenorphine, and oxycodone at baseline and follow-up; UDS will also test for other substances including cocaine, amphetamines, and THC.
California prescription drug monitoring database (CURES) | Baseline, weeks 1-14, post-treatment (week 15), and 2 months from week 15
  Opioid and benzodiazepine prescriptions (including dose) will be corroborated by review of the CURES system.
Anxiety Sensitivity Index-3 (change) | Baseline, bi-weekly during weeks 1-14, post-treatment (week 15), and 2 months from week 15
  The ASI-3 measures anxiety sensitivity (cognitive misappraisals of anxiety as being harmful, or "fear of fear."). ASI-3 will be given frequently throughout treatment to establish temporal precedence needed to assess for possible mediation of treatment outcomes.
Pain Catastrophizing Scale (change) | Baseline, bi-weekly during weeks 1-14, post-treatment (week 15), and 2 months from week 15
  The Pain Catastrophizing Scale will be used as a secondary outcome associated with opioid prescription use and will be given frequently throughout treatment to establish temporal precedence needed to assess for possible mediation of treatment outcomes.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - UCLA Health MPTF Toluca Lake Primary Care, Burbank, California
  - UCLA Integrated Substance Abuse Programs, Los Angeles, California
  - UCLA Family Health Center, Santa Monica, California

IPD SHARING:
Plan to Share IPD: Yes
Per NIH guidelines, we provide a data sharing plan for the study. The study MPIs will collaborate with the NIH to finalize public use dataset procedures, ensure that the rights and privacy of all individual research participants are protected at all times, and that Protected Personal Health Information (PHI) is protected as required by law and approved by the study IRBs. We will share our data via National Institute of Health Data Archive (NDA). NDA links data across research projects through its Global Unique Identifier (GUID) and Data Dictionary technology. We will use these technologies to submit data to NDA.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Wolitzky-Taylor K, Mooney LJ, Otto MW, Metts A, Parsons EM, Hanano M, Ram R. Augmenting the efficacy of benzodiazepine taper with telehealth-delivered cognitive behavioral therapy for anxiety disorders in patients using prescription opioids: A pilot randomized controlled trial. Contemp Clin Trials. 2023 Oct;133:107334. doi: 10.1016/j.cct.2023.107334. Epub 2023 Sep 18. PMID 37730196